CLINICAL TRIAL: NCT02105337
Title: A Pilot Study: Does Tegaderm Placement on Eyes to Prevent Lagophthalmos Affect Visual Evoked Potentials Data Latency and Amplitude
Brief Title: Tegaderm and Visual Evoked Potentials
Status: Terminated | Type: Observational
Why Stopped: PI leaving institution
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Anesthesia, Division of Neuroanesthesia, Rutgers, The State University of New Jersey
Other Study IDs: 2013002781
Record Dates: First submitted 2014-01-15; First posted 2014-04-07 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2014-09

CONDITIONS: Tumor of Pituitary and Suprasellar Region
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tegaderm placement: all pts will have tegaderm placed prior to goggles for VEP

SUMMARY:
The purpose of this study is to determine if a clear barrier placed over the eyes has any effect on goggle monitoring. When a patient has general anesthesia they lose the ability to blink and their eyes may dry. They may also lose the ability to keep their eyes fully closed. The anesthesiologist takes several steps to prevent injury to the eyes. First the eyes will be lubricated with ointment and the eyelids will be held in a closed position by the use of a clear barrier. During pituitary surgery it is the routine practice to perform many types of monitoring. One type of monitoring is to stimulate your eyes with a light. This helps your surgeon protect the nerve supply to your eyes. The light is supplied by a pair of goggles placed over your eyes during surgery.

To help achieve our objective, the investigators are asking patients who are undergoing pituitary surgery to give us permission to record two sets of numbers form the monitoring device once prior to the application of the clear barrier and the second after the barrier is applied. This will be done when the patient is already asleep and will not be aware this is happening.

DETAILED DESCRIPTION:
Corneal injury is the most frequent ocular complication during general anesthesia as the patient does not have the ability to blink or keep their eyes completely closed. Lagophthalmos is defined as the inability to close the eyelids completely. Blinking covers the eye with a thin layer of tear fluid, thereby promoting a moist environment necessary for the cells of the exterior part of the eye. The tears also flush out foreign bodies and wash them away. This is crucial to maintain lubrication and proper eye health. If this process is impaired, as in lagophthalmos, the eye can suffer abrasions and infections. Lagophthalmos leads to corneal drying and ulceration. Several strategies are widely used to try and prevent corneal abrasions, although there is a paucity of recent studies to support one method over another. If a patient is to receive general anesthesia the common practice is to lubricate the eyes and tape them closed.

One of the ways to prevent lagophthalmos is to use tegaderm. A tegaderm is a thin transparent barrier customarily used to protect wounds and catheter sites. The tegaderm has several advantages including breathability and conformity to skin. In the operating room it is place over the patients' eyelids to keep the eyes closed and prevent injury.

During surgical removal of a pituitary adenoma, conduction in the anterior visual pathways is monitored by continuous recording of visual evoked potentials (VEP). The VEP tests the function of the visual pathway from the retina to the occipital cortex. It measures the conduction of the visual pathways from the optic nerve, optic chiasm, and optic radiations to the occipital cortex. This method is performed by the application of special goggles over the eyes. These goggles placed over the tegaderm are noninvasive and have an embedded flashing diode for delivery of visual stimuli. Changes of the occipital EEG (as recorded intraoperatively on a computer program by a neurophysiology technician) can be observed under stimulation of light in attempt to localize structures or possible damage of those structures in the primary visual pathway. This is helpful to the neurosurgeon who aims to avoid compression and injury to the optic nerve.

These goggles have been used routinely over years for visual pathway monitoring during pituitary tumor resection. Nevertheless there is a question if the application of tegaderm affects VEP monitoring. By measuring visual evoked potentials before and after tegaderm placement, we hope to determine if there is a change in evoked potential data due to placement of tegaderm. On other words, we will be able to identify if tegaderm placement affects visual evoked potential data reliability.

Experimental Plan:

The investigators will approach all patients over the age of 18 undergoing transsphenoidal pituitary tumor resection with visual evoke potential monitoring.The plan is to include 40 patients here at University Hospital. If patients are agreeable all subjects will have their VEP measured before and after routine tegaderm application. Visual evoked potential monitoring will be conducted as routinely done by the neurophysiology technician. Data will be collected from neurophysiologist report and then analyzed for latency and amplitude before and after tegaderm application. As a matter of routine, the full monitoring report becomes a component of the patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

>18 years of age -

Exclusion Criteria:

no history of diabetic retinopathy not currently pregnant

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: undergoing transsphenoidal pituitary tumor resection with visual evoked potential
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
change in latency of VEP | 1 minute
  Visual evoked potential data in terms of latency and amplitude will be compared before and after tegaderm placement and statistically analyzed. We expect to make pilot preliminary conclusion if tegaderm application affects visual evoked potential monitoring in term of latency and amplitude of the data.

SECONDARY OUTCOMES:
Change in amplitude of VEP | 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Pisklakov, MD, Principal Investigator — Rutgers/SUNJ
Locations (1):
- University Hospital, Newark, New Jersey, United States